CLINICAL TRIAL: NCT06486129
Title: Long-term Myocardial Effects of Noninvasive Ventilation in Patients With Obesity Hypoventilation Syndrome
Brief Title: Myocardial Effects of NIV in OHS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pavol Jozef Safarik University (Other)
Responsible Party: Principal Investigator, Pavol Pobeha, Pavol Pobeha, MD, PhD (Principal investigator), Pavol Jozef Safarik University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEGA 1/0220/17
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Failure Chronic; Obesity Hypoventilation Syndrome; Obstructive Sleep Apnea; Cardiac Output, Low
Keywords: Respiratory Failure; Obesity Hypoventilation Syndrome; Obstructive Sleep Apnea; Cardiac Output; stroke volume
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Sleep Apnea, Obstructive; Cardiac Output, Low; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Clinically stable patients with OHS and severe hypercapnia during the daytime, referred to the tertiary clinic for the initiation of long-term NIV to alleviate chronic respiratory failure were consecutively enrolled to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obesity hypoventilation syndrome patients treated with BPAP (NIV) therapy (Experimental): Clinically stable patients with OHS and severe hypercapnia during the daytime, referred to the tertiary clinic for the initiation of long-term NIV to alleviate chronic respiratory failure were consecutively enrolled to the study
  Interventions: Procedure: Noninvasive ventilation volume targetted

INTERVENTIONS:
Procedure: Noninvasive ventilation volume targetted — he aim of the present study was to evaluate the long-term effects of volume-targeted bilevel-positive airway pressure ventilation (BiPAP) on cardiac parameters and myocardial biomarkers in patients with OHS

SUMMARY:
Chronic effects of noninvasive ventilation on myocardial function in patients with obesity hypoventilation syndrome (OHS) are scarcely understood. The aim of the present study was to evaluate the long-term effects of volume-targeted bilevel-positive airway pressure ventilation (BiPAP) on cardiac parameters and myocardial biomarkers in patients with OHS.

DETAILED DESCRIPTION:
Chronic effects of non- invasive ventilation on myocardial function in patients with obesity hypoventilation syndrome (OHS) are scarcely understood. The aim of the present study was to evaluate the long-term effects of volume-targeted bilevel-positive airway pressure ventilation (BiPAP) on cardiac parameters and myocardial biomarkers in patients with OHS. Clinically stable patients with OHS referred to the tertiary centre for the initiation of long-term BiPAP therapy were consecutively enrolled in the study. At baseline, all participants underwent overnight cardiorespiratory polygraphy. BiPAP therapy using volume-targeted spontaneous/timed mode delivered via an oro-nasal mask was initiated. Beat-to-beat noninvasive monitoring by impedance cardiography was used to assess heart function at baseline and after 3 and 12 months of BiPAP use. Serum troponin 1, N-Terminal Pro-B-Type Natriuretic Peptide (NTProBNP), tumor necrosis factor-alpha (TNF-α), and interleukin-6 (IL-6) were monitored. Potential risks and benefits comprise haemodynamic effects of NIV on cardiovascular parameters including cardiac output and stroke volume. The study started 06/2016 and enrolment was finalized in October 2018. The study was funded by grants from the Slovak Research and Development Agency under contract No. APVV-16-0158, and VEGA 1/0220/17 and 1/0393/22 of the Ministry of Education, Slovakia. The main investigator is Pavol Pobeha, MD, PhD, co author is Ivana Paranicova, MD, PhD and the corresponding author (study coordinator prof. Ruzena Tkacova, MD, PhD)

ELIGIBILITY:
Inclusion Criteria:

- Clinically stable patients with OHS and chronic severe hypercapnia

Exclusion Criteria:

* inability to provide written informed consent
* neuromuscular diseases
* chest wall diseases
* metabolic diseases
* acute respiratory tract infection
* chronic obstructive pulmonary disease (COPD)
* systolic LV failure as evidenced by LV ejection fraction<45% on echocardiography

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Impedance cardiography measured cardiac output | 12 months
  Impedance cardiography measured cardiac output before and after effective treatment of respiratory failure

SECONDARY OUTCOMES:
Impedance cardiography measured stroke volume | 12 months
  Impedance cardiography measured stroke volume before and after effective treatment of

CONTACTS AND LOCATIONS:
Locations (1):
- Department of respiratory medicine and tuberculosis, Pavol Jozef Safarik University, Medical Faculty and L. Pasteur University Hospital In Kosice, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided
On request

REFERENCES:
- [Background] Pobeha P, Paranicova I, Trojova I, Tkacova R, Joppa P. Acute hemodynamic effects of non-invasive ventilation in patients with obesity hypoventilation syndrome. Bratisl Lek Listy. 2021;122(4):248-250. doi: 10.4149/BLL_2021_040. PMID 33729816